CLINICAL TRIAL: NCT06095570
Title: The Study of Ciprofol for the Suppression of Cardiovascular Responses to Tracheal
Brief Title: The Study of Ciprofol for the Suppression of Cardiovascular Responses to Tracheal Intubation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Hainan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RM20220701
Record Dates: First submitted 2023-09-30; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Intubation, Intratracheal; Adverse Effects
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; remimazolam; 4-methylbenzenesulfonic acid; Injections

STUDY DESIGN:
Intervention Model Description: Group C: Ciprofol + sufentanil + rocuronium bromide Group R: Remimazolam+ sufentanil + rocuronium bromide
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: People who were unaware of the experiment helped to randomize the groups and inject the test drug according to the groups, and the patients who participated in the experiment as well as the doctors were unaware of the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Experimental): Ciprofol + sufentanil + rocuronium bromide
  Interventions: Drug: Ciprofol
- Group R (Active Comparator): Remimazolam+ sufentanil + rocuronium bromide
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Ciprofol — For induction of anesthesia, an experimental dose of ciprofol was given, and when the patient lost consciousness and the Modified Observer's Alertness/Sedation scale(MOAA/S score) was less than 1, then intravenous sufentanil and rocuronium bromide were administered, and tracheal intubation was performed 3 minutes later
  Other Names: Ciprofol injection
  Arms: Group C
Drug: Remimazolam — For induction of anesthesia, an experimental dose of remimazolam was given, and when the patient lost consciousness and the Modified Observer's Alertness/Sedation scale(MOAA/S score) was less than 1, then intravenous sufentanil and rocuronium bromide were administered, and tracheal intubation was performed 3 minutes later
  Other Names: Remimazolam Tosylate for Injection
  Arms: Group R

SUMMARY:
Preliminary studies have illuminated the promising nature of ciprofol, indicating its enhanced safety spectrum, superior potency, and a diminished likelihood of experiencing injection-related discomfort. Venturing deeper, this research embarked on an ambitious quest to measure the 95% effective volume of ciprofol for induction of general anesthesia by a modified sequential method and juxtapose the 95% effective volume dosage of ciprofol against a corresponding dose of remimazolam during the initiation of general anesthesia. The study delved into diverse anesthetic protocols, meticulously scrutinizing the safety and efficacy credentials of ciprofol. The ultimate vision was to pave a robust foundation for the sophisticated and judicious utilization of ciprofol in clinical landscapes.

DETAILED DESCRIPTION:
During general anesthesia induction, tracheal intubation is a significant procedure that can cause cardiovascular fluctuations due to the stimulation of tracheal receptors. This can lead to complications such as imbalances in vital organ oxygen supply, especially in patients with cardiovascular and cerebrovascular disorders, potentially resulting in cardiac arrest. As the demand for anesthetics rises in clinical settings, some, due to extreme side effects, have been phased out, reducing the available options.

Propofol, a common anesthetic, is effective and quick but has drawbacks like injection pain and risks associated with long-term use. In contrast, ciprofol, a new class I intravenous anesthetic, is emerging as a potentially better alternative. Early research indicates that ciprofol might have a broader safety margin than propofol and offers benefits like rapid recovery and lower chances of injection pain.

Exhaustive studies on the precise dosage of ciprofol for surgical applications are scarce and comparisons between ciprofol and remimazolam are rarely reported in the literature. This research aims to bridge this knowledge gap, exploring the best dosage for tracheal intubation sedation, and ensuring patients get the most effective and safest anesthetic care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing surgery with a single-lumen endotracheal tube placed under general anesthesia;
2. American Society of Anesthesiologists(ASA grade) I or II;
3. Age 18~65 years old;
4. Body mass index (BMI) 18 to 28 kg/m2;
5. Mallampati airway classification grade I or II;
6. Acceptance of this experiment and signing of informed consent.

Exclusion Criteria:

1. Patients with a history of alcoholism, allergy to any component of the product;
2. Patients with severe heart, lung and brain vital organ diseases, such as acute heart attack, cerebral infarction, asthma, chronic obstructive pulmonary disease and other medical history;
3. Serious liver and kidney function abnormalities or combined serious endocrine dysfunction, such as hypertension (systolic blood pressure ≥ 160 mmHg, diastolic blood pressure ≥ 110 mmHg, HR ≥ 110 beats/min), diabetes mellitus, hyperthyroidism, hypothyroidism and so on;
4. Difficult airway (mouth opening less than 3 cross fingers, those with Mallampati score grade III or IV, difficulty in vocal valve exposure, difficulty in tracheal intubation, unsuccessful in one attempt); oropharyngeal and cervical deformities or history of previous tracheotomy;
5. Neuropsychiatric abnormalities, communication and comprehension deficits exist;
6. History of long-term sedative and analgesic medications, drug and opioid addiction, and heart rate control medications (e.g., beta blockers, alpha agonists, calcium channel blockers); and
7. Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-07-23 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Heart Rate(HR) | Intravenous ciprofol up to 3 minutes after tracheal intubation
  Heart rate monitored with Dash4000 equipment
Mean Arterial Pressure(MAP) | Intravenous ciprofol up to 3 minutes after tracheal intubation
  Heart rate monitored with Dash4000 equipment

SECONDARY OUTCOMES:
Bispectral Index(BIS) | Intravenous ciprofol up to 3 minutes after tracheal intubation
  Monitored woth Bispectral Index Vista. BIS ranges from 0-100, with 100 representing full wakefulness and 0 representing complete cortical electroencephalogram(EEG) suppression; the smaller the value, the deeper the depth of sedation Mild sedation is BIS 65-85, and deep sedation is BIS 40-60, with primitive EEG bursts of suppression when BIS < 40.
Peripheral Oxygen Saturation(SPO2) | Intravenous ciprofol up to 3 minutes after tracheal intubation
  Monitored with Dash4000 equipment
Rate of respiratory inhibition,Injection pain,Hypotension,Allergy,Bradycardia,Muscle tremor,Postoperative nausea and vomiting | Intravenous ciprofol to leave resuscitation
  Referring to the standards in ciprofol's Phase III trial, the adverse reactions were defined as follows: (1) hypoxemia (oxygen saturation < 90% for > 30 s); (2) bradycardia (HR < 45/min for > 30 s); (3) hypotension (systolic BP decreased by 30% from the baseline value for > 2 min); and (4) pain at the injection site during ciprofol administration, evaluated by a study-blinded investigator using a 4-point verbal rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hu Sun, Study Chair — The Second Affiliated Hospital of Hainan Medical University, Hai Kou, China; Min Liao, Study Director — The Second Affiliated Hospital of Hainan Medical University, Hai Kou, China; Xiaoru Wu, Principal Investigator — The Second Affiliated Hospital of Hainan Medical University, Hai Kou, China; Jianing Hu, Principal Investigator — The Second Affiliated Hospital of Hainan Medical University, Hai Kou, China; Xingzhou Lin, Principal Investigator — The Second Affiliated Hospital of Hainan Medical University, Hai Kou, China; Tangyuanmeng Zhao, Principal Investigator — West China Hospital
Locations (1):
- The Second Affiliated Hospital of Hainan Medical University, Hai Kou, China, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: No
Non-disclosure of raw data is not necessary

REFERENCES:
- [Background] El-Shmaa NS, El-Baradey GF. The efficacy of labetalol vs dexmedetomidine for attenuation of hemodynamic stress response to laryngoscopy and endotracheal intubation. J Clin Anesth. 2016 Jun;31:267-73. doi: 10.1016/j.jclinane.2016.01.037. Epub 2016 Apr 18. PMID 27185725
- [Background] Kayhan Z, Aldemir D, Mutlu H, Ogus E. Which is responsible for the haemodynamic response due to laryngoscopy and endotracheal intubation? Catecholamines, vasopressin or angiotensin? Eur J Anaesthesiol. 2005 Oct;22(10):780-5. doi: 10.1017/s0265021505001298. PMID 16211744
- [Background] Higgs A, McGrath BA, Goddard C, Rangasami J, Suntharalingam G, Gale R, Cook TM; Difficult Airway Society; Intensive Care Society; Faculty of Intensive Care Medicine; Royal College of Anaesthetists. Guidelines for the management of tracheal intubation in critically ill adults. Br J Anaesth. 2018 Feb;120(2):323-352. doi: 10.1016/j.bja.2017.10.021. Epub 2017 Nov 26. PMID 29406182
- [Background] Xue FS, Xu YC, Liu Y, Yang QY, Liao X, Liu HP, Zhang YM, Liu JH, Luo MP. Different small-dose sufentanil blunting cardiovascular responses to laryngoscopy and intubation in children: a randomized, double-blind comparison. Br J Anaesth. 2008 May;100(5):717-23. doi: 10.1093/bja/aen032. Epub 2008 Mar 5. PMID 18325887
- [Background] Weisenberg M, Sessler DI, Tavdi M, Gleb M, Ezri T, Dalton JE, Protianov M, Zimlichmann R. Dose-dependent hemodynamic effects of propofol induction following brotizolam premedication in hypertensive patients taking angiotensin-converting enzyme inhibitors. J Clin Anesth. 2010 May;22(3):190-5. doi: 10.1016/j.jclinane.2009.07.008. PMID 20400005
- [Background] Sneyd JR, Absalom AR, Barends CRM, Jones JB. Hypotension during propofol sedation for colonoscopy: a retrospective exploratory analysis and meta-analysis. Br J Anaesth. 2022 Apr;128(4):610-622. doi: 10.1016/j.bja.2021.10.044. Epub 2021 Dec 13. PMID 34916051
- [Background] Hemphill S, McMenamin L, Bellamy MC, Hopkins PM. Propofol infusion syndrome: a structured literature review and analysis of published case reports. Br J Anaesth. 2019 Apr;122(4):448-459. doi: 10.1016/j.bja.2018.12.025. Epub 2019 Feb 6. PMID 30857601
- [Background] Qin L, Ren L, Wan S, Liu G, Luo X, Liu Z, Li F, Yu Y, Liu J, Wei Y. Design, Synthesis, and Evaluation of Novel 2,6-Disubstituted Phenol Derivatives as General Anesthetics. J Med Chem. 2017 May 11;60(9):3606-3617. doi: 10.1021/acs.jmedchem.7b00254. Epub 2017 Apr 28. PMID 28430430
- [Background] Bian Y, Zhang H, Ma S, Jiao Y, Yan P, Liu X, Ma S, Xiong Y, Gu Z, Yu Z, Huang C, Miao L. Mass balance, pharmacokinetics and pharmacodynamics of intravenous HSK3486, a novel anaesthetic, administered to healthy subjects. Br J Clin Pharmacol. 2021 Jan;87(1):93-105. doi: 10.1111/bcp.14363. Epub 2020 Aug 3. PMID 32415708
- [Derived] Liao M, Wu XR, Hu JN, Lin XZ, Zhao TY, Sun H. Comparative effective dose of ciprofol and propofol in suppressing cardiovascular responses to tracheal intubation. Sci Rep. 2025 Jan 13;15(1):1822. doi: 10.1038/s41598-025-85968-2. PMID 39805976